CLINICAL TRIAL: NCT01753011
Title: Prospective, Observational Study: Can Pelvic Floor Ultrasound Help to Optimize TOT (Transobturator Tape) Positioning?
Brief Title: Urethral Length and TOT (Transobturator Tape) Positioning
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital, Frauenfeld (Other)
Responsible Party: Principal Investigator, Prof. Dr. Volker Viereck, Prof. Dr. Volker Viereck, Cantonal Hospital, Frauenfeld
Other Study IDs: TOT 1/2-Rule
Record Dates: First submitted 2012-12-17; First posted 2012-12-19 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress urinary Incontinence; Transobturator sling; TOT
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Stress Urinary Incontinence: Stress Urinary Incontinence

SUMMARY:
This is a prospective, observational, multicenter study of women with surgically-correctable stress urinary incontinence who undergo a TOT-sling operative procedure.

DETAILED DESCRIPTION:
This is a prospective, observational, multicenter study of women with surgically-correctable stress urinary incontinence who undergo a TOT-sling operative procedure. Data will be collected from preoperative urogynecological testing and medical histories. Outcome data will be collected 1-3 days and 6 months after procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has objective demonstrable signs of stress urinary incontinence (SUI), including patients with intrinsic sphincter deficiency (ISD). Objective testing includes: standing stress test, urodynamics evaluation, or pad test.
2. Patient is age 18 or older.
3. Patient agrees to participate in the study, including completion of all study-related procedures and evaluations, and documents this agreement by signing the Institutional Review Board (IRB)/Ethic commission (EC)-approved informed consent.
4. Patient is able to fill in all questionnaires (on judgement of investigator)

Exclusion Criteria:

1. Patient has an associated or suspected neurological disease.
2. Patient has an active lesion or present injury to perineum or urethra.
3. Patient has a urethral obstruction.
4. Patient has significant pelvic organ prolapse (Grade III/IV) requiring surgical treatment.
5. Patient currently has an urinary tract infection.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes women with surgically-corrected stress urinary incontinence who undergo a TOT operative procedure.
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2007-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Cure rate | 6 months postoperative
  The primary outcome of the TOT procedure will be assessed using a combination of objective and subjective criteria. Patients with a negative stress test, a negative 1-h pad test (less than 2 g) and the degree of subjective suffering improving to over 90% (VAS score of 0-1) at 6 months follow-up evaluation are classified as cured. All other patients are classified as treatment failure even if one aspect shows marked improvement from the preoperative condition.

SECONDARY OUTCOMES:
Urethral length | Preoperative
  Urethral length will be measured by pelvic floor sonography.
Linear urethral dorsocaudal movement (LUDM) | Preoperative
  Linear urethral dorsocaudal movement (LUDM) will be assessed by pelvic floor sonography.
Urethral tape position | 1-3 days and 6 months postoperative
  The position of the TOT along the urethra will be determined by pelvic floor sonography and expressed as percentage of urethral length.
Distance between tape and longitudinal smooth muscle (LSM) complex | 1-3 days and 6 months postoperative
  To characterize the location of the TOT, the shortest distance between the tape and the longitudinal smooth muscle (LSM) complex of the urethra will be measured by pelvic floor sonography.
Urodynamic testing | Preoperative
  Urodynamic testing will be performed only for patients undergoing recurrent incontinence surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Volker Viereck, Prof. Dr., Principal Investigator — Cantonal Hospital, Frauenfeld
Locations (2):
- Department of Gynecology and Obstetrics, Lutheran Hospital Hagen-Haspe, Hagen, Germany
- Blasenzentrum, Cantonal Hospital, Frauenfeld, Thurgau, Switzerland